CLINICAL TRIAL: NCT07241923
Title: A Phase I, Single-Center, Randomized, Double-Blind, Placebo-Controlled, Single-Ascending-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SYH2070 Injection in Healthy Subjects
Brief Title: A Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SYH2070 Injection
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYH2070-001
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Healthy Subjects (HS)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYH2070 experimental group (Experimental): Subjects in experimental groups will receive a single subcutaneous injection of SYH2070 injection on Day 1.
  Interventions: Drug: SYH2070 injection
- Placebo group (Placebo Comparator): Subjects in placebo groups will receive a single subcutaneous injection of placebo on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SYH2070 injection — subcutaneous injection
  Arms: SYH2070 experimental group
Drug: Placebo — subcutaneous injection
  Arms: Placebo group

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single ascending dose (SAD) study of SYH2070 injection when administered subcutaneously to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide informed consent before the trial, fully understand its content, procedures, and potential adverse reactions, and voluntarily sign the written ICF;
2. Sex: Male or female;
3. Age: 18-60 years (inclusive);
4. Body mass index (BMI) in the range of 19 to 30 kg•m^2 [BMI = weight/height^2 (kg•m^2)] (inclusive), with a weight of no less than 50 kg for males (inclusive) and no less than 45 kg for females (inclusive);
5. Fasting serum TG ≥150 mg/dL (1.7 mmol/L) and ≤ 500 mg/dL (5.6 mmol/L), and LDL-C ≥70 mg/dL (1.8 mmol/L) and < 190 mg/dL (4.9 mmol/L) during the screening and baseline periods;
6. Subjects must maintain stable die, exercise, and other lifestyle habits from 4 weeks prior to screening until the end of the study, with no planned changes to diet, exercise or weight loss programs;
7. Subjects must be able to communicate well with the investigator and can complete the study according to the protocol requirements.

Exclusion Criteria:

1. History of severe allergic diseases or allergic constitution (≥ 3 drug or food allergies), or known history of allergy to the investigational drug components (N-acetylgalactosamine, sodium hydroxide, phosphoric acid) or oligonucleotide drugs;
2. Use of antibody drugs and/or oligonucleotide drugs targeting PCSK9/ANGPTL3/ApoC-III within 12 months prior to screening;
3. Current and/or history of clinically significant medical conditions, including but not limited to circulatory, hematological or hematopoietic, respiratory, endocrine, urinary, digestive system diseases, neurological or psychiatric disorders, infections, tumors, severe trauma, or any other disease that should be excluded or may interfere with the interpretation of the study results, as judged by the investigator;
4. History of major surgery within 6 months prior to screening, or are scheduled to undergo major surgery during the course of the study;
5. History of bariatric surgery within 12 months prior to screening;
6. Have clinically significant abnormalities in vital signs, physical examination, electrocardiogram, and laboratory tests (excluding lipid parameters);
7. Estimated glomerular filtration rate (eGFR) <90 mL/min/1.73 m^2 at screening;
8. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (TBIL), gamma-glutamyl transferase (GGT), or alkaline phosphatase (ALP) >1.5× upper limit of normal (ULN) at screening (one retest allowed within 1 week);
9. Prolonged QT / QTc interval at screening or baseline (QTcF > 450 ms);
10. Positive result for any of HBsAg, HCV antibody, syphilis antibody, and HIV antibody;
11. Blood loss or donation >200 mL within 3 months prior to screening (excluding menstruation for females), and/or platelet donation within 2 weeks;
12. Use of any drugs, health supplements, vitamins, or dietary supplements known to affect lipid metabolism within the longer of either: (a) 28 days prior to dosing; (b) 7 half-lives of the drug; (3) the duration of the agent's pharmacological effect, including but not limited to statins, fish oil, high-purity omega-3, prescription-dose niacin, fibrates, or anti-estrogen therapy;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with Adverse Events as Assessed by CTCAE v5.0 | Pre-dose and multiple time points no less than 85 days

SECONDARY OUTCOMES:
The serum TG level after dosing SYH2070 injection | Pre-dose and multiple timepoints no less than 85 days
The serum LDL-C level after dosing SYH2070 injection | Pre-dose and multiple timepoints no less than 85 days
Plasma Maximum concentration (Cmax) | Pre-dose and multiple timepoints up to 4 days
Time to maximum concentration (Tmax) | Pre-dose and multiple timepoints up to 4 days
Area under the concentration-time curve from 0 to the collection time t (AUC0-t) | Pre-dose and multiple timepoints up to 4 days
Half-Life (t1/2) | Pre-dose and multiple timepoints up to 4 days
Area under the concentration-time curve from 0 to infinity (AUC0-∞) | Pre-dose and multiple timepoints up to 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials Information Group, Shijiazhuang, Hebei, China